CLINICAL TRIAL: NCT00716391
Title: Open Label Randomized, Multi-centre Phase III Trial of TPF Plus Concomitant Treatment With Cisplatin and Radiotherapy Versus Concomitant Cetuximab and Radiotherapy in Locally Advanced, Unresectable Head and Neck Cancer.
Brief Title: TPF Plus Cisplatin and Radiotherapy vs TPF Plus Cetuximab and Radiotherapy to Treat Head and Neck Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Grupo Español de Tratamiento de Tumores de Cabeza y Cuello (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTCC-2007-01
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2019-05-24 (Actual); Status verified 2019-05

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Radiotherapy; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Active Comparator): TPF plus concomitant treatment with cisplatin and conventional radiotherapy.
  Interventions: Other: TPF, radiotherapy and cisplatin.
- Group B (Experimental): TPF plus concomitant treatment with cetuximab and conventional radiotherapy
  Interventions: Other: TPF, radiotherapy and cetuximab.

INTERVENTIONS:
Other: TPF, radiotherapy and cisplatin. — 3 cycles of: cisplatin: 75 mg/m2, i.v., 1 hour, once daily docetaxel: 75 mg/m2, i.v., 1 hour, once daily 5-fluorouracil: 750 mg/m2, i.v., 24 hours, 5 days Radiotherapy: 70Gy, divided into daily doses of 2 Gray (total days: 35) Cisplatin: 100 mg/m2, i.v., 1 hour, 3 days
  Other Names: TPF plus radiotherapy and cisplatin
  Arms: Group A
Other: TPF, radiotherapy and cetuximab. — 3 cycles of: cisplatin: 75 mg/m2, i.v., 1 hour, once daily docetaxel: 75 mg/m2, i.v., 1 hour, once daily 5-fluorouracil: 750 mg/m2, i.v., 24 hours, 5 days Radiotherapy: 70Gy, divided into daily doses of 2 Gray (total days: 35) Cetuximab: 400 mg/m2, i.v, 2 hours, 1 day Cetuximab: 250 mg/m2, i.v, 1 hour, 7 days
  Other Names: TPF plus radiotherapy and cetuximab
  Arms: Group B

SUMMARY:
An Open Label Randomized, Multi-Centre Phase III Trial of TPF Chemotherapy Plus Concomitant Treatment With Cisplatin and Conventional Radiotherapy Versus TPF Chemotherapy Plus Concomitant Cetuximab and Conventional Radiotherapy in Locally Advanced, Unresectable Head and Neck Cancer.

DETAILED DESCRIPTION:
This study is being sponsored by a cooperative medical group.

ELIGIBILITY:
Inclusion Criteria:

1. Before the beginning of protocol's specific procedures, the informed consent has to be obtained.
2. Locally advanced cancer of head and neck (oral cavity, oropharynx, larynx and hypopharynx) stage III-IV, without evidence of metastasis.
3. The tumor must be considered to be non-operable according to the criteria of the Northern California Oncology Group. The reason of non-surgical resection will be annotated in the CRF.

   Criteria of non-surgical resection according to the NCOG:

   3.1.Technically not resectable (includes: evidence of mediastinal dissemination; fixed tumor to the clavicle, base of the cranium or cervical vertebrae; affectation of the nasopharynx).

   3.2.Medical criteria based on a low surgical curability. 3.3.Medical contraindication for the surgery.
4. Epidermoid carcinoma histologically demonstrated
5. Measurable disease according to the RECIST criteria .
6. Men or women with age between 18 and 70 years, both inclusive.
7. Functional condition index according to ECOG scale:0-1
8. Patients in medical conditions to be able to receive treatment with TPF induction followed by normofractionated radiotherapy with cetuximab or cisplatin.
9. Patients with adequate hematologic function: neutrophils superior or equal to 2 x 109, platelets superior or equal to 100 x 109, hemoglobin superior or equal to 10 g/dl.
10. Adequate hepatic function: bilirubin lower or equal to 1 x top normal Limit, GOT and GPT lower or equal to 2,5 Top Normal Limit , alkaline phosphatase < 5 Top Normal Limit.
11. Adequate renal function: creatinin <1,4 mg/dl (120 µmol/l); if the values are > 1,4 mg/dl, the clearance of creatinin will have to be > 60 ml/min (real or calculated for Cockcroft-Gault's method).
12. Calcium lower or equal to 1,25 x top normal limit.
13. Adequate nutritional condition: loss of weight <20% with relation to the theoretical weight and albumin superior or equal to 35 g/L.
14. Patients must be accessible for the treatment and the follow-up.

Exclusion Criteria:

1. Metastatic disease
2. Surgical treatment, previous radiotherapy and/or chemotherapy for the study disease.
3. Other tumor locations in head and neck that are not oral cavity, oropharynx, larynx, hypopharynx.
4. Other stages that are not III or IVM0.
5. Other previous and / or synchronic squamous carcinoma.
6. Diagnosis of another neoplasia in the last 5 years, excepting carcinoma in situ of uterine neck and/or a cutaneous carcinoma basocellular properly treated.
7. Active infection(at needs endovenous antibiotics), including active tuberculosis and diagnosed HIV.
8. Not controlled hypertension defined as arterial systolic tension superior or equal to 180 mm Hg and / or diastolic arterial tension superior or equal to 130 mm Hg baseline.
9. Pregnancy(absence must be confirmed with the test of beta-HCG) or period of lactation.
10. Immunity systemic treatment, chronic and concomitant, or hormonal treatment of the cancer.
11. Other antineoplastic concomitant treatments.
12. Coronary clinically significant arteriopathy or precedents of myocardial infarction in the last 12 months or high risk of not controlled arrhythmia or cardiac not controlled insufficiency.
13. Pulmonary obstructive chronic disease that had needed 3 or more hospitalizations in the last 12 months.
14. Active non controlled peptic ulcer.
15. Presence of a psychological or medical disease that could prevent to accomplish the study by the patient or to grant his/her signature in the informed consent form.
16. Known drugs abuse (with the exception of excessive consumption of alcohol)
17. Known allergic reaction to some of the components of the treatment of the study.
18. Previous treatment with monoclonal antibodies or other transduction of the sign inhibitors or treatment directed against the EGFR.
19. Any experimental treatment in 30 days before the entry in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 519 (Actual)
Dates: Start 2008-07-07 (Actual); Primary Completion 2017-07-18 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Global survival | Up to 89 months
  The time from the start of induction chemotherapy with TPF to death due to any cause or to the last check-up in the case of living patients

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 89 months
  The response rate (CR + PR) measured using the RECIST 1.0 method.
Progression free-survival (PFS) | Up to 89 months
  Time to progression as the time since the start date of treatment with TPF induction chemotherapy until the time when DP occurred or death occurred due to any cause.
Time to loco-regional control of disease | Up to 89 months
  As permanent and complete resolution of the disease in terms of its initial site and lymph nodes (T and N). If the disease lasted (regardless of size), the tumor recurred, or a second tumor appeared in the field RT, it will be recorded as a therapeutic failure.
Satisfaction with treatment. Analysis of QoL in both treatment arms. | Up to 89 months
  EORTC QoL questionnaires: C30 version 3.0 and QLQ-H&N35 module

CONTACTS AND LOCATIONS:
Overall Officials: Juan J Cruz, Professor, Principal Investigator — University of Salamanca; Ricardo Hitt, MD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (39):
- Spain (39):
  - Hospital Puerta del Mar, Almería, Almería
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Durán i Reynals, Hospitalet de Ll., Barcelona
  - Hospital de Manresa, Manresa, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Son Dureta, Palma de Mallorca, Mallorca
  - Hospital Son Llàtzer, Palma de Mallorca, Mallorca
  - Hospital de Sagunto, Sagunto, Valencia
  - Hospital general Universitario, Alicante
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital Clínic i Provincial de Barcelona, Barcelona
  - Hospital de Basurto, Bilbao
  - Hospital General Yagüe, Burgos
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Dr. Trueta (ICO Girona), Girona
  - Oncogranada, Granada
  - H. Virgen de las Nieves, Granada
  - Hospital General de Jaén, Jaén
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Xeral Calde, Lugo
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Clínica Quirón, Madrid
  - Fundación Jiménez Díaz, Madrid
  - Hospital Gregorio Marañon, Madrid
  - Hospital La Paz, Madrid
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Clínico de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Hospital Arnau de Vilanova, Valencia
  - Hospital General Universitario, Valencia
  - Hospital La Fe, Valencia
  - Hospital Xeral Cies, Vigo
  - Hospital de Meixoeiro, Vigo
  - Hospital Provincial de Zamora, Zamora
  - Hospital Clínico Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- See also: This site would like to expose the activities of the group and at the same time serve as an information and communication tool of this pathology for professionals and patients. — http://www.ttccgrupo.org/

DOCUMENTS (2):
  • Study Protocol (2012-04-30): https://cdn.clinicaltrials.gov/large-docs/91/NCT00716391/Prot_000.pdf
  • Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT00716391/SAP_001.pdf